CLINICAL TRIAL: NCT01112592
Title: The Ability of Neutrophils From Patients With Recurrent Infections to Produce Neutrophil Extracellular Traps (NET).
Brief Title: NETs Formation in Patients With Recurrent Pyogenic Infections (NETS)
Acronym: NETs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Max Planck Institute for Infection Biology (Other)
Responsible Party: Sponsor
Other Study IDs: MMC-10156-09CTIL
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2012-03

CONDITIONS: Pyogenic Infections
Keywords: NETs; Infections; Neutrophil function
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
We aim to study if pathological NETs formation could be the underlying pathology among patients with recurrent infections and a normal screening of the immune system.

DETAILED DESCRIPTION:
Our laboratory at Meir Medical Center, Kfar Saba, is the country's main center for neutrophil function, and serves about 80% of Israel's population. Patients are referred subsequent to recurrent, persistent, or unusual infections and after completing preliminary screening of the immune system and ruling out a humoral, cellular or complement immune deficiency. Initial workup includes chemotaxis, superoxide production (SOP), and bactericidal activity (BA). Based on test findings, further evaluation for a qualitative phagocytic disorder is conducted. Overall, impairment of phagocytic activity is found in about 33% (impaired chemotaxis in 16%, SOP in 6%, and BA in 24%). In the other 67%, no impairment of the immune function is found that can explain their tendency for recurrent pyogenic infections.

In 2004 a novel function of the neutrophil was identified: formation of neutrophil extracellular traps (NETs). Apparently, neutrophils are able to extrude part of their cellular contents in the form of DNA, histones and proteases, to form extra cellular NETS that trap and kill bacterial pathogens without the need for phagocytosis. We aim to study if pathological NETs formation could be the underlying pathology among these patients with recurrent infections and a normal screening of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent, persistent, or unusual infections
* Referred for Neutrophil Functions

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients are referred subsequent to recurrent, persistent, or unusual infections and after completing preliminary screening of the immune system and ruling out a humoral, cellular or complement immune deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Measure NET formation in patients with recurrent infections | One year

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Wolach, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel